CLINICAL TRIAL: NCT05185700
Title: Post Covid 19 Syndrome
Brief Title: Symptoms ,Signs and Complications That Appear After Infection With Covid 19 Virus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Kamal Darwish, Specialist , chest department and tuberculosis, Assiut University
Other Study IDs: post covid 19 syndrome
Record Dates: First submitted 2022-01-09; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: post covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: post covid 19 symtoms — observation

SUMMARY:
1. Raise awareness for persistent post-COVID syndrome (PPCS).
2. Rising tide of physical and psychological disabilities that have been described in post-COVID patients.

DETAILED DESCRIPTION:
Since SARS-CoV-2 infection was recognised in late 2019, the academic and clinical emphasis has been on respiratory manifestations .

Post-COVID syndrome appears to be a multisystem disease, occurring even after a relatively mild acute illness. Increasing evidence exists for direct multiorgan effects, and indirect effects on other organ systems and disease processes, such as cardiovascular diseases and cancers, through changes in healthcare delivery and patient behaviors . So, the long term effects of covid-19 on individuals and health systems are becoming clear, investigation across organ systems is urgently needed. Long covid, or post-covid syndrome, is not one condition, and is defined by the National Institute for Health and Care Excellence (NICE) as "signs and symptoms that develop during or after an infection consistent with covid-19 which continue for more than 12 weeks and are not explained by an alternative diagnosis . NICE guidelines recommend referral to post-covid syndrome assessment clinics if post covid symptoms persist for 6-12 weeks . Pre-existing conditions and risk factors are predictors of acute covid-19 outcomes (such as admission to the intensive care unit and mortality, but the epidemiology of postcovid syndrome has been less well defined . Because of the unclear medium and long term pathophysiology across organ systems. When post-covid syndrome clinics are established, characterization of the epidemiology of the disease will help with appropriate diagnosis, care, public health interventions and policy, and resource planning. So, further research is highly indicated.

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed as covid-19.
* Presence of post covid-19 symptoms.

Exclusion Criteria:

* Patient refusal.
* Patient less than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective study will be conducted on 175 patients who were previously diagnosed as covid-19. A written consent will be obtained from the patient or from his first degree-relative.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Identifying post covid -19 respiratory manifestations. | 1 year
  detection of respiratory symptoms and signs appears within 6 months after infection with covid 19

SECONDARY OUTCOMES:
identifying other post covid -19 manifestations. | 1 year
  detection of extra respiratory manifestions of covid 19 infection to improve outcome of post covid 19 patients

CONTACTS AND LOCATIONS:
Overall Officials: Rafaat T El-Sokry, professor, Study Director — assuit university hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Puntmann VO, Carerj ML, Wieters I, Fahim M, Arendt C, Hoffmann J, Shchendrygina A, Escher F, Vasa-Nicotera M, Zeiher AM, Vehreschild M, Nagel E. Outcomes of Cardiovascular Magnetic Resonance Imaging in Patients Recently Recovered From Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Nov 1;5(11):1265-1273. doi: 10.1001/jamacardio.2020.3557. PMID 32730619
- [Background] Tabary M, Khanmohammadi S, Araghi F, Dadkhahfar S, Tavangar SM. Pathologic features of COVID-19: A concise review. Pathol Res Pract. 2020 Sep;216(9):153097. doi: 10.1016/j.prp.2020.153097. Epub 2020 Jul 4. PMID 32825963
- [Background] Alqahtani SA, Schattenberg JM. Liver injury in COVID-19: The current evidence. United European Gastroenterol J. 2020 Jun;8(5):509-519. doi: 10.1177/2050640620924157. PMID 32450787
- [Background] Somasundaram NP, Ranathunga I, Ratnasamy V, Wijewickrama PSA, Dissanayake HA, Yogendranathan N, Gamage KKK, de Silva NL, Sumanatilleke M, Katulanda P, Grossman AB. The Impact of SARS-Cov-2 Virus Infection on the Endocrine System. J Endocr Soc. 2020 Jul 2;4(8):bvaa082. doi: 10.1210/jendso/bvaa082. eCollection 2020 Aug 1. PMID 32728654
- [Background] Farouk SS, Fiaccadori E, Cravedi P, Campbell KN. COVID-19 and the kidney: what we think we know so far and what we don't. J Nephrol. 2020 Dec;33(6):1213-1218. doi: 10.1007/s40620-020-00789-y. Epub 2020 Jul 20. PMID 32691342
- [Background] Ball S, Banerjee A, Berry C, Boyle JR, Bray B, Bradlow W, Chaudhry A, Crawley R, Danesh J, Denniston A, Falter F, Figueroa JD, Hall C, Hemingway H, Jefferson E, Johnson T, King G, Lee KK, McKean P, Mason S, Mills NL, Pearson E, Pirmohamed M, Poon MTC, Priedon R, Shah A, Sofat R, Sterne JAC, Strachan FE, Sudlow CLM, Szarka Z, Whiteley W, Wyatt M; CVD-COVID-UK Consortium. Monitoring indirect impact of COVID-19 pandemic on services for cardiovascular diseases in the UK. Heart. 2020 Dec;106(24):1890-1897. doi: 10.1136/heartjnl-2020-317870. Epub 2020 Oct 5. PMID 33020224
- [Background] Lai AG, Pasea L, Banerjee A, Hall G, Denaxas S, Chang WH, Katsoulis M, Williams B, Pillay D, Noursadeghi M, Linch D, Hughes D, Forster MD, Turnbull C, Fitzpatrick NK, Boyd K, Foster GR, Enver T, Nafilyan V, Humberstone B, Neal RD, Cooper M, Jones M, Pritchard-Jones K, Sullivan R, Davie C, Lawler M, Hemingway H. Estimated impact of the COVID-19 pandemic on cancer services and excess 1-year mortality in people with cancer and multimorbidity: near real-time data on cancer care, cancer deaths and a population-based cohort study. BMJ Open. 2020 Nov 17;10(11):e043828. doi: 10.1136/bmjopen-2020-043828. PMID 33203640
- [Background] Katsoulis M, Gomes M, Lai AG, Henry A, Denaxas S, Lagiou P, Nafilyan V, Humberstone B, Banerjee A, Hemingway H, Lumbers RT. Estimating the Effect of Reduced Attendance at Emergency Departments for Suspected Cardiac Conditions on Cardiac Mortality During the COVID-19 Pandemic. Circ Cardiovasc Qual Outcomes. 2021 Jan;14(1):e007085. doi: 10.1161/CIRCOUTCOMES.120.007085. Epub 2020 Dec 20. No abstract available. PMID 33342219
- [Background] Greenhalgh T, Knight M, A'Court C, Buxton M, Husain L. Management of post-acute covid-19 in primary care. BMJ. 2020 Aug 11;370:m3026. doi: 10.1136/bmj.m3026. No abstract available. PMID 32784198
- See also: Related Info — https://apps.who.int/iris/handle/10665/331446
- See also: Related Info — http://directorsblog.nih.gov/tag/post-covid-syndrome
- See also: Related Info — https://evidence.nihr.ac.uk/themedreview/living-with-covid19/